CLINICAL TRIAL: NCT06646432
Title: Treatment of Gingival Recession by Tunnel Technique Using Connective Tissue Graft With or Without Injectable Platelet Rich Fibrin: A Randomized Controlled Clinical Trial
Brief Title: Treatment of Gingival Recession With Tunnel Technique Using Connective Tissue Graft and Injectable Platelet Rich Fibrin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 486/2022
Record Dates: First submitted 2024-10-03; First posted 2024-10-17 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Gingival Recession
Keywords: Tunneling; Gingival recession; Injectable platelet rich fibrin; Minimally invasive periodontology
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group: tunnel with connective tissue graft and injectable platelet rich fibrin (Experimental): Tunneling will be performed at the recession defect sites with insertion of palatal connective tissue graft taken from the patient hard palate inside the prepared tunnel. The graft will be soaked ,before insertion inside the tunnel, in injectable platelet rich fibrin ,prepared from patient own blood for 15 minutes. The tunnel with the soaked graft inside will be advanced coronally.
  Interventions: Procedure: Tunnel with connective tissue graft and injectable platelet rich fibrin
- Control group: tunnel with connective tissue graft only (Active Comparator): Tunnel preparation will be made in the recession defect sites with insertion of palatal connective tissue graft from the patient hard palate. The tunnel with the graft will be advanced coronally.
  Interventions: Procedure: Tunnel with connective tissue graft only

INTERVENTIONS:
Procedure: Tunnel with connective tissue graft and injectable platelet rich fibrin — Tunnel with connective tissue graft and injectable platelet rich fibrin
  Arms: Test group: tunnel with connective tissue graft and injectable platelet rich fibrin
Procedure: Tunnel with connective tissue graft only — Tunnel technique with connective tossue graft only without injectable platelet rich fibrin
  Arms: Control group: tunnel with connective tissue graft only

SUMMARY:
Gingival recession is a common periodontal problem. Consequences include teeth sensitivity, poor esthetics and impaired oral hygiene access. Mild cases are managed by optimizing oral hygiene measures, correction of any causative factor such as faulty tooth brushing, improper dental restoration or denture clasp. Prescription of desensitization products such as specific tooth gels or mouth washes can manage the sensitivity problem. Deeper recession defects need to be addressed by surgical procedures. Coronally advanced flap with connective tissue graft is the gold standard procedure. However, it has some drawbacks due to the need for papillary incisions and vertical incisions in some cases. Within the era of minimally invasive periodontology, tunnel technique with connective tissue graft showed results comparable to coronally advanced flap with connective tissue graft but with some limitations. Addition of another agent may enhance the results of tunnel technique. Injectable platelet rich fibrin is known for its content of growth factors and effects on soft tissue healing. Aim: The study aim is to compare the surgical management of gingival recession with tunnel technique using connective tissue graft and injectable platelet rich fibrin to tunnel with connective graft without injectable platelet rich fibrin.

Methodology: 30 patients with miller class I or II gingival recession will be enrolled. 15 in the test group (Tunnel+ CTG+ i-PRF) and 15 in control group (Tunnel+ CTG). Clinical evaluation at 6 months

DETAILED DESCRIPTION:
30 patients with miller class I/II gingival recession will be enrolled in this study.

15 patients will be treated using tunnel technique and palatal connective tissue graft inserted and sutured under the prepared tunnel after being soaked in injectable platelet rich fibrin for 15 minutes. The tunnel with the underlying graft will be advanced coronally. (Test Group) The other 15 patients will be treated the same way as in the first group but without soaking the graft in injectable platelet rich fibrin. (Control Group) Clinical parameters will be evaluated at baseline and 6 months follow-up except post-operative pain which will be assessed after 10 days. Histologic examination of small piece of the graft will be done to assess if there is true saturation of growth factors inside the graft.

ELIGIBILITY:
Inclusion Criteria:

* More than 21 years old
* Systemically healthy
* Presence of Miller class I/II gingival recession
* Presence of identifiable CEJ

Exclusion Criteria:

* Smoking
* Systemic disease that contraindicates surgical procedures.
* Poor compliance with oral hygiene measures
* Necrotizing gingival conditions
* Ongoing active periodontitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Recession depth | 6 months after the surgery
  it will be recorded as the distance between the CEJ and gingival margin-measurements were performed at the mid-buccal aspect of the teeth, by manual probe and were rounded up to the nearest millimeter.
Keratinized tissue height | 6 months
  It will be measured from the mucogingival junction to the gingival margin-measurements were performed at the mid-buccal aspect of the teeth, by manual probe and were rounded up to the nearest millimeter.
Gingival thickness | 6 months
  It will be measured at a mid-buccal location 1 mm apical to the probing depth level with an spreader. It will be pierced, perpendicularly to the mucosal surface, through the soft tissue with light pressure until a hard surface is felt. The silicone disk stop will then be placed in tight contact with the soft tissue surface. Penetration depth will be measured.

SECONDARY OUTCOMES:
Post operative pain | 10 days
  It will be measured by Visual analog Scale (VAS) with records from 0 to 10 with 0 means no pain and 10 means very severe pain. The patient will report the degree he experienced pain and choose a score from VAS.
Recession width | 6 months
  It will be measured horizontally between the borders of the recession at the level of Cemento-enamel Junction.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelnasser Elrefaey, Study Chair — Suez Canal University; Shaimaa Morsy, Study Director — Suez Canal University
Locations (1):
- Faculty of dentistry, Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No